CLINICAL TRIAL: NCT05175846
Title: Observational Study of Immunological and INFLAMmatory BiomarkErs in COVID-19 Naïve and Infected Participants and Severity of Disease
Brief Title: INFLAMmatory BiomarkErs in COVID-19 Participants and Severity of Disease
Acronym: INFLAME COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trinitas Global, LLC (Industry)
Collaborators: AccessDx Laboratories, Houston, TX (Unknown)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2021-12-28; First posted 2022-01-04 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: COVID-19, inflammatory biomarkers
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma collected for testing of inflammatory biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal volunteers: Participants with negative COVID-19 test
- COVID-19: Participants with positive COVID-19 test and severe symptoms of disease

SUMMARY:
Observational Study of the Association of Immunological and Inflammatory Biomarkers in COVID-19 Naïve and Infected Participants and Severity of Disease. Thirty naive and 30 COVID positive participants will have a blood sample taken after informed consent and be assessed for COVID symptoms according to WHO classification. Participants will be followed monthly for 6 months. At each contact, participants will be assessed for COVID symptoms and progress since the previous visit.

DETAILED DESCRIPTION:
This is an observational study of participants who are being or have been tested for COVID-19. Participants with or without COVID-19 will be entered into one of two groups for Stage 1 and one of three groups for Stage 2.

Stage 1:

* Group 1: Participants whose COVID-19 test is negative and who do not have symptoms of COVID-19 disease.
* Group 2: Participants whose COVID-19 test is positive and who have Severe or Critical symptoms of COVID-19 disease.

Stage 2:

* Group 1: Participants whose COVID-19 test is negative and who do not have symptoms of COVID-19 disease.
* Group 2: Participants whose COVID-19 test is positive and who have Mild or Moderate symptoms of COVID-19 disease.
* Group 3: Participants whose COVID-19 test is positive and who have Severe or Critical symptoms of COVID-19 disease.

During Stage 1, Group 1 participants will be matched to Group 2 subjects as follows: Age: 18-64 and >65; Race: Caucasian, Latino, African American, other; Sex: Male or Female Each participant will be assigned a study number. The study case report form (CRF) will record the participants initials, age and study number. Participants will have blood drawn for biomarkers. All samples will be identified using the participants age and study number. Blood volume will be approximately ten milliliters to yield at least four 1 ml serum aliquots. Serum will be frozen at -80ºF and stored. Batch shipments of the serum will occur during the study and sent to AccessDx Laboratory in Houston TX. Laboratory procedures for AccessDx are presented in Appendices B and C. AccessDx will perform the following biomarker tests on the serum: Interleukins 1B, 6, 8,10, 22; CRP; Ferritin; Interferon-ꝩ; MIP 1α and 1β; TNF; VEGF A, B, C.

Participants will be followed for up to 6 months and have monthly calls from the study staff. As much as possible, the participant will be contacted by the same study member at each follow-up visit. If agreed with the participant, information about the participants status may be collected on email or text. Participants will be asked specific questions and their responses recorded on a paper CRF. At enrollment and at each follow-up call, the participant's severity of COVID-19 disease will be categorized based on WHO Interim guidance 27 May 2020 as follows:

* Mild cases are marked by the onset of symptoms such as fever, cough, fatigue, shortness of breath, headache, diarrhea, and so forth, without evidence of viral pneumonia or hypoxia.
* Moderate cases include clinical signs of pneumonia (fever, cough, dyspnea, fast breathing) but no signs of severe pneumonia, including SpO2 ≥ 90% on room air.
* Severe cases demonstrate clinical signs of pneumonia (fever, cough, dyspnea, fast breathing) plus one of the following: respiratory rate > 30 breaths/min; severe respiratory distress; or SpO2 < 90% on room air.
* Critical cases present symptoms such as acute respiratory distress syndrome (ARDS), sepsis and/or septic shock A participant's engagement in the study will be approximately 6 months. Recruitment is expected to last 6 months. It is expected that the total study for Stage 1 will be one year. The duration of Stage 2 will not be determined until results from Stage 1 are available. The number of investigator sites for Stage 1 is expected to be up to 3 and for Stage 2, up to 50.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (IC) within 4 days of COVID-19 test.
2. Age 18 or older
3. COVID-19 test

Group 1: negative COVID-19 test Group 2: positive COVID-19 test with Severe or Critical symptoms of disease (per WHO Guidance).

Exclusion Criteria:

1. Any autoimmune disease or immune-modulator therapy.
2. Mild or Moderate symptoms of COVID-19 disease (per WHO Guidance).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants at least 18 years of age who do not have autoimmune disease or are not taking immune-modulator therapy and may or may not have a positive COVID-19 test will be entered into one of two groups for Stage 1 of the study. (Stage 2 is TBD).
  * Group 1: Participants whose COVID-19 test is negative and who do not have symptoms of COVID-19 disease.
  * Group 2: Participants whose COVID-19 test is positive and who have Severe or Critical symptoms of COVID-19 disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
To identify immunological and inflammatory biomarkers in participants with and without COVID-19 that may predict a participant's potential risk for severity of disease. | 30 days
  Correlation of biomarkers at baseline with severity of COVID-19 disease at baseline and on Day 30 according to WHO classification of COVID-19 symptoms

SECONDARY OUTCOMES:
To correlate the biomarkers at baseline with the duration of symptoms up to six months in participants who develop COVID-19. | 6 months
  Duration and severity of symptoms of COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Monteleone, MD, Principal Investigator — Saint Francis Family Medicine Residency Program, Wilmington, Delaware
Locations (1):
- St Francis Hospital, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No